CLINICAL TRIAL: NCT04465656
Title: Registry of the Evolution of Diagnosed and/or Hospitalized Patients for Pulmonary Embolism During the Covid-19 Pandemic: Retrospective and Prospective Multicentric Study.
Brief Title: Registry of the Evolution of Diagnosed and/or Hospitalized Patients for Pulmonary Embolism During the Covid-19 Pandemic
Acronym: COVID-EP
Status: Completed | Type: Observational
Sponsor: Hospital St. Joseph, Marseille, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-05-01
Record Dates: First submitted 2020-06-30; First posted 2020-07-10 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — Serologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- [PCR-COVID 19-Pos] group: Having a microbiological diagnosis confirming COVID-19 infection (ie positive RT-PCR on nasopharyngeal swab) and/or clinical/CT signs
- [PCR-COVID 19-Neg] group: Having a microbiological diagnosis confirming the absence of COVID-19 infection (ie negative RT-PCR on nasopharyngeal swab) and absence of clinical /CT signs
  Interventions: Diagnostic Test: Serology test for COVID-19
- [PCR-COVID 19-Neg & Sero-COVID 19-Pos] group: * Having a microbiological diagnosis confirming the absence of COVID-19 infection (ie negative RT-PCR on nasopharyngeal swab) and absence of clinical /CT signs
  * Having been tested positive in a serological test for COVID-19 at M3
- [PCR-COVID 19-Neg & Sero-COVID 19-Neg] group: * Having a microbiological diagnosis confirming the absence of COVID-19 infection (ie negative RT-PCR on nasopharyngeal swab) and absence of clinical /CT signs
  * Having been tested negative in a serological test for COVID-19 at M3

INTERVENTIONS:
Diagnostic Test: Serology test for COVID-19 — In order to secondarily confirm the COVID-19 status of initially negative COVID-19 patients (by RT-PCR), a serology test will be performed in two parts:
  1. ELISA test
  2. Rapid Diagnostic tests (only if ELISA test is positive)
  Groups: [PCR-COVID 19-Neg] group

SUMMARY:
The purpose of the study COVID-EP is to classify all the complications occurring after the diagnosis of pulmonary embolism in patients tested initially COVID-19 positive and negative by RT-PCR (on nasopharyngeal sample) during the peak of the pandemic in France (April 2020). The patients will be followed for 1 year in order to provide clinical and paraclinical data not yet published in the literature. In order to secondarily confirm the COVID-19 status of initially negative COVID-19 patients (by RT-PCR), a serology test will be performed. The collected complications will then be compared between each of the 3 following groups: [PCR-COVID 19-Neg & Sero-COVID 19-Neg] versus [PCR-COVID 19-Neg & Sero-COVID 19-Pos] versus [PCR-COVID 19-Pos].

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years,
* Diagnosed for pulmonary embolism between April 1st and April 30th, 2020; (treated by ambulatory care or hospitalized),
* Having given free and informed written consent,
* Being affiliated with or benefiting from a social security scheme.

Exclusion Criteria:

* Subject to a measure for the protection of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient diagnosed and / or hospitalized for PE in April 2020 (the COVID-19 pandemic peak)
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2022-09-08 (Actual)

PRIMARY OUTCOMES:
% of patients for each group presenting the occurrence of PE complications defined by the occurrence of at least ONE of the following events up to 6 months after PE diagnosis. | 6 months after PE diagnosis
  PE complications :
  * Chronic interstitial pathology, or
  * Recurrence of PE, or
  * Pulmonary hypertension, or
  * Death.

SECONDARY OUTCOMES:
% of patients for each group and subgroup presenting the occurrence of PE complications defined by the occurrence of at least ONE of the following events up to 12 months after PE diagnosis. | 12 months after PE diagnosis
  PE complications :
  * Chronic interstitial pathology, or
  * Recurrence of PE, or
  * Pulmonary hypertension, or
  * Death.
% of patients in each group presenting the occurrence of each of the following events at each follow-up (3 months, 6 months and 12 months after PE diagnosis). | 3, 6 and 12 months after PE diagnosis
  PE complications :
  * Chronic interstitial pathology, or
  * Recurrence of PE, or
  * Pulmonary hypertension, or
  * Death.
% of patients diagnosed COVID - at M0 by RT-PCR on nasopharyngeal swab and diagnosed COVID + by serology 3 months after PE diagnosis | 3 months after PE diagnosis
Effectiveness of the different category of treatments used in all patients and in the groups: % of occurrence of PE complications for each categories of treatments | 12 months after PE diagnosis
  Category of treatments:
  * Heparin + AVK
  * Heparin + DOAC
  PE complication :
  * Chronic interstitial pathology, or
  * Recurrence of PE, or
  * Pulmonary hypertension, or
  * Death.
Effectiveness of the different category of treatments used in all patients and in the groups: % of patients with occurrence of bleeding complications for each categories of treatments | 12 months after PE diagnosis
  Category of treatments:
  * Heparin + AVK
  * Heparin + DOAC
  Bleeding complications: classification 1-2-3-5 according to BARC
Effectiveness of the different category of treatments used in all patients and in the groups: % of patients with no occurrence of complications for each categories of treatments | 12 months after PE diagnosis
  Category of treatments:
  * Heparin + AVK
  * Heparin + DOAC
Effectiveness of the different category of treatments used in all patients and in the groups: duration of Heparin treatment (number of day) | 12 months after PE diagnosis
  Category of treatments:
  * Heparin + AVK
  * Heparin + DOAC

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Saint Joseph Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No